CLINICAL TRIAL: NCT06031480
Title: Study of Combination Treatment Using Anlotinib and TQB2450 in Patients With Advanced Hepatocellular Carcinoma Who Failed Prior Immune Checkpoint Inhibitor Therapies: a Single Arm, Multicenter Clinical Trial
Brief Title: Anlotinib and TQB2450 in Advanced Hepatocellular Carcinoma After Failure of Prior Immune Checkpoint Inhibitors
Acronym: FAITH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2023297
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib+TQB2450 (Experimental)
  Interventions: Drug: Anlotinib and TQB2450

INTERVENTIONS:
Drug: Anlotinib and TQB2450 — Anlotinib: 10mg PO, QD, D1-14, Q3W; TQB2450: 1200 mg, IV, D1, Q3W.
  Anlotinib and TQB2450 will be administered until the disease progression, intolerable toxicity, death, withdrawal of consent.

SUMMARY:
This is an multi-center, single arm, exploratory study to evaluate the efficacy and safety of anlitinib combined with TQB2450 in patients with advanced hepatocellular carcinoma （HCC）who failed prior immune checkpoint inhibitor therapies.

ELIGIBILITY:
Inclusion Criteria:

* The participants must be required to sign an informed consent
* Hepatocellular carcinoma patients confirmed by pathological or cytological examination, or who meet the clinical diagnostic criteria of the "Guidelines for the Diagnosis and Treatment of primary hepatocellular carcinoma" (2022)
* At least one measurable lesion (RECIST 1.1)
* Chinese Liver Cancer Staging (CNLC): CNLC-IIa, IIb, IIIa, IIIb (BCLC-B and C) that are not suitable for local treatment (TACE, HAIC, etc.) or that have progressed after local treatment
* The previous treatment plan for patients before enrollment was a standard treatment plan containing immune checkpoint inhibitors, and patients with progression or intolerance were evaluated based on the RECIST v1.1 standard
* Child-Pugh Score, Class A or better B
* ECOG performance status 0 or 1
* Adequate organ function
* Life expectancy of at least 3 months

Exclusion Criteria:

* Patients who have received local treatment (including TACE, ablation, HAIC, radiotherapy) and are less than 1 month after enrollment
* Patients who have received ≥ 2 treatments with immune checkpoint inhibitor regimens
* Adverse events above level 1(NCI-CTCAE v5.0) caused by any previous treatment that have not returned to ≤ level 1 (excluding hair loss); Patients with previous severe immune-related AEs requiring permanent cessation of immunotherapy
* Pregnant or lactating wome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR, RECIST v1.1) | 24 months
  ORR is defined as the proportion of subjects with complete response (CR) or partial response (PR) to study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, Shanghai Municipality, China